CLINICAL TRIAL: NCT01243112
Title: Onset and Duration of Effect of Lidocaine, Bupivacaine, and Lidocaine/Bupivacaine Mixture With Epinephrine.
Brief Title: Effectiveness Study of Different Local Anesthetic Mixtures
Acronym: CA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scott and White Hospital & Clinic (Other)
Responsible Party: Principal Investigator, James Collins, MD, Scott and White Hospital & Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 090520
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Results first posted 2011-12-02 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Epinephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lidocaine w/ Epi (Experimental): 0.2ml 1% Lidocaine with Epinephrine (1:100,000)
  Interventions: Drug: 1% Lidocaine with Epinephrine (1:100,000)
- Bupivacaine with epi (Experimental): 0.2 ml 0.25% Bupivacaine with epinephrine (1:200,000)
  Interventions: Drug: 0.25% Bupivacaine with Epinephrine (1:200,000)
- Low dose Lido and Bupi w/ Epi (Experimental): 0.2ml 0.5% Lidocaine + 0.125% Bupivacaine with Epinephrine (1:150,000)
  Interventions: Drug: 0.5% Lidocaine, 0.125 Bupivacaine, and epi (1:150,000)
- High Dose Lido and Bupi with epi (Experimental): 0.2ml 1% Lidocaine + 0.25% Bupivacaine with Epinephrine (1:150,000)
  Interventions: Drug: 1% Lidocaine, 0.5% Bupivacaine, and epinephrine (1:150,000)

INTERVENTIONS:
Drug: 1% Lidocaine with Epinephrine (1:100,000) — 0.2ml Intradermal injection once.
  Arms: Lidocaine w/ Epi
Drug: 0.25% Bupivacaine with Epinephrine (1:200,000) — 0.2ml Intradermal injection once.
  Arms: Bupivacaine with epi
Drug: 0.5% Lidocaine, 0.125 Bupivacaine, and epi (1:150,000) — 0.2ml Intradermal injection once.
  Arms: Low dose Lido and Bupi w/ Epi
Drug: 1% Lidocaine, 0.5% Bupivacaine, and epinephrine (1:150,000) — 0.2ml Intradermal injection once.
  Arms: High Dose Lido and Bupi with epi

SUMMARY:
Purpose and Background The purpose of this research study is to investigate the benefits of mixing lidocaine and bupivacaine for numbing the skin. Lidocaine and bupivacaine are two commonly used medications to numb the skin for minor procedures. Lidocaine has a faster onset. Bupivacaine has a longer duration. They are often combined with epinephrine to increase the length of action. These medications are used to control pain at the time of the operation and to decrease discomfort immediately afterward. Participating in the study involves injection of local anesthetic containing lidocaine, bupivacaine, and lidocaine and bupivacain with epinephrine at 4 sites on the forearm. Your participation will potentially improve the administration of these medications in persons undergoing a variety of procedures. You will be one of approximately 25 healthy volunteer subjects in this research study.

DETAILED DESCRIPTION:
Procedures

During your participation the following procedures will be completed:

* You will be asked to read over and sign this consent form, if you choose to participate
* You will be asked demographic information and your medical history will be obtained
* If you are eligible to participate, the palm side of your forearm will be marked for the location of the treatments
* Four small injections will be made into the palm side of your forearms with the local anesthetic mixtures (you will not know which injection is used at each of the four injection sites)
* A small needle will be used for pinprick sensation to determine when numbness begins and ends

Length of Study and Number of Visits This study begins at the time the medications are injected and is completed when sensation has completely returned. The study will last between 6 and 12 hours. During this time, you may perform low intensity tasks including reading, typing, and writing. You must remain in the study location as the sites will frequently be examined.

Exclusions

You should not participate in this study if any of the following apply to you:

* You are pregnant
* You have an allergy to lidocaine or bupivacaine
* You have a history of heart disease (including a prior heart attack, heart dysfunction, or heart failure)

There may be other criteria that you have to meet to be eligible for this study. The study team can discuss these with you to determine whether you qualify.

Discomfort and Risks Risks associated with the injections include temporary discomfort at the injection site and possible infection. It is also possible that you have an allergic reaction or side effect to the medications that are being used.

Benefits There is no direct benefit to you for participating in this study. Your participation will potentially improve the administration of these medications in persons undergoing a variety of procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60

Exclusion Criteria:

* Pregnancy
* allergy to local anesthetics
* history of heart disease or diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Collins, MD, Principal Investigator — Scott and White Healthcare; Raman C Mahabir, MD, Study Director — Scott and White Healthcare
Locations (1):
- Scott & White, Temple, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by hospital mailing list with 25 subjects enrolled over May 2010 until September 2010.
Groups:
- Study Group: 0.2 ml 1% Lidocaine with Epinephrine (1:100,000), 0.2 ml 0.25% Bupivacaine with Epinephrine (1:200,000) 0.2 ml 0.5% Lidocaine and 0.125% Bupivacaine with Epinephrine Epinephrine (1:150,000) 2 ml of 1% Lidocaine and 0.25% Bupivacaine with Epinephrine (1:150,000)
Period: Overall Study
Arm/Group | Study Group
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Length of Action
Description: The time from onset of local anesthesia until cessation of effect by sensation of sharp measured in 15 minute increments.
Time Frame: Up to 12 hours
Population: A calculation was made to power the study appropriately to determine a difference of 5 minutes based on previous studies which did not include the use of epinephrine.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Study Group
Number analyzed (Participants) | 25
minutes
  1% Lidocaine With Epinephrine | 6.63 (1.85)
  0.25% Bupivacaine With Epinephrine | 7.02 (1.46)
  0.5% Lidocaine and 0.125% Bupivacaine With Epineph | 7.48 (1.76)
  1% Lidocaine and 0.25% Bupivacaine With Epinephrin | 7.16 (1.60)
Statistical Analysis 1: Comparison: Study Group; Null Hypothesis is that no difference would be measured between treatment arms; Test type: Superiority or Other; p = 0.359, ANOVA

2. Primary Outcome: Onset of Action
Description: Time from infusion of local anesthetic to loss of sensation to sharp.
Time Frame: Up to 5 minutes
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Study Group
Number analyzed (Participants) | 25
second
  1% Lidocaine With Epinephrine | 29 (49)
  0.25% Bupivacaine With Epinephrine | 19 (41)
  0.5% Lidocaine and 0.125% Bupivacaine With Epineph | 26 (46)
  1% Lidocaine and 0.25% Bupivacaine With Epinephrin | 12 (30)
Statistical Analysis 1: Comparison: Study Group; Test type: Superiority or Other; p = 0.490, ANOVA

ADVERSE EVENTS:
Time Frame: 7/24/10 to 8/28/10
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes